CLINICAL TRIAL: NCT04444141
Title: A Multicenter, Open-label, Phase Ib/II Study of AK104, a PD-1/CTLA-4 Bispecific Antibody, in Subjects With Relapsed or Refractory Peripheral T Cell Lymphoma
Brief Title: A Study of PD-1/CTLA-4 Bispecific AK104 in Relapsed or Refractory Peripheral T-cell Lymphoma
Status: Terminated | Phase: Phase 1 / Phase 2 | Type: Interventional
Why Stopped: Due to difficuty of erollment and consideration of clinical guideline,The sponsor decided to stop study.
Sponsor: Akeso (Industry)
Collaborators: Akeso Pharmaceuticals, Inc. (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: AK104-203
Record Dates: First submitted 2020-06-21; First posted 2020-06-23 (Actual); Last update posted 2022-10-19 (Actual); Status verified 2022-10

CONDITIONS: Peripheral T-cell Lymphoma
Keywords: Anti-PD-1; Anti-CTLA-4; Bispecific
MeSH Terms: conditions — Lymphoma, T-Cell, Peripheral

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- AK104 (Experimental): AK104 450mg IV every 2 weeks (Q2W)
  Interventions: Biological: AK104

INTERVENTIONS:
Biological: AK104 — The subjects will receive AK104 till disease progression or for a maximum of 24 months.

SUMMARY:
The purpose of this study is to evaluate the efficacy and safety of AK104，an anti- PD-1 and CTLA-4 bispecific antibody, in subjects with relapsed or refractory peripheral T cell lymphoma. The subject will receive AK104 450mg Q2W until unacceptable toxicity, confirmed disease progression, withdrawal of consent, or for a maximum of 24 months.

ELIGIBILITY:
Inclusion Criteria:

* Patients with histologically or cytologically confirmed advanced Peripheral T-cell lymphoma.
* Relapsed or refractory disease after at least 1 prior systemic treatment for the primary malignancy and not a candidate for other curative treatments.
* Eastern Cooperative Oncology Group (ECOG) physical fitness score is 0 or 1.
* Adequate organ functions
* Effective methods of contraception.
* Ability to provide written informed consent and to be compliant with the schedule of protocol assessments.

Exclusion Criteria:

* Patients diagnosed as adult T cell lymphoma / leukemia (ATLL).
* Any prior exposure to PD-1/PD-L1、CTLA-4 targeting agents.
* Previous allogeneic stem cell transplant within 3 months prior to enrolment, active graft vs host disease (GVHD), or requiring transplant-related immunosuppression.
* Serious systemic infections or local infections during the 2 months before screening.
* History of cancer in 5 years before screening., including solid tumors and hematological malignancies (except basal cell and in situ squamous cell carcinomas of the skin that have been excised and resolved).
* Have a known allergy or hypersensitivity to any biologic therapy at screening that would pose an unacceptable risk to the subject if participating in this study.
* Has enrolled in any other trials during 3 months prior to screening or concurrently enrolled in any other trials.
* Received allogeneic organ transplantation or allogeneic hematopoietic stem cell transplantation.
* Subjects who received immunomodulatory drugs in 4 weeks before screening, including thymosin, interferon and interleukin, et al.
* Patients who received radiotherapy, chemotherapy, targeted therapy (except TKI), immunotherapy within 4 weeks before screening, and patients who received TKI drugs within 2 weeks before screening.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 6 (Actual)
Dates: Start 2020-05-15 (Actual); Primary Completion 2022-09-30 (Actual); Study Completion 2022-09-30 (Actual)

PRIMARY OUTCOMES:
Objective response rate (ORR) | Up to 2 years
  Objective response is defined as the proportion of subjects with confirmed CR or PR according to the Lugano 2014 classification for lymphoma, assessed by the investigator.

SECONDARY OUTCOMES:
Progression-free survival (PFS) | Up to 2 years
  Progression-free survival is defined as the time from the start of treatment with AK104 until the first documentation of disease progression or death due to any cause, whichever occurs first.
Disease control rate (DCR) | Up to 2 years
  The DCR is defined as the proportion of subjects with CR, PR, or SD according to the Lugano 2014 classification for lymphoma.
Duration of response (DoR) | Up to 2 years
  Duration of response is defined as the duration from the first documentation of objective response to the first documented disease progression or death due to any cause, whichever occurs first.
Number of subjects experiencing adverse events (AEs) | From the time of informed consent signed through 90 days after the last dose of AK104
  The incidence and severity of adverse events, containing clinically significant abnormal laboratory tests, vital signs and electrocardiogram (ECG) results.
Number of subjects who develop detectable anti-drug antibodies (ADAs) | From first dose of AK104 through 90 days after last dose of AK104
  The immunogenicity of AK104 will be assessed by summarizing the number of subjects who develop detectable antidrug antibodies (ADAs).
Observed concentrations of AK104 | From first dose of AK104 through 90 days after last dose of AK104
  The endpoints for assessment of PK of AK104 include serum concentrations of AK104 at different timepoints after AK104 administration.

CONTACTS AND LOCATIONS:
Overall Officials: Yuqin Song, MD, Principal Investigator — Peking University Cancer Hospital & Institute; Jun Zhu, MD, Principal Investigator — Peking University Cancer Hospital & Institute
Locations (1):
- Beijing Cancer Hospital, Beijing, Beiing, China